CLINICAL TRIAL: NCT06245473
Title: Characterization of Metabolomic Fingerprints in Patients With Hepatic Encephalopathy
Brief Title: Metobolomics in the Characterisation of HE
Acronym: METABO-EH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220279
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: Hepatic encephalopathy; Cirrhosis; Metabolomics
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 6-mL tube for metabolomic analysis during a blood test scheduled as part of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample — During the blood test planned as part of the care an additional blood tube with a volume of 6mL will be takeń in an EDTA tube.

SUMMARY:
Hepatic encephalopathy is (HE) defined by the neurological and/or neuropsychological symptoms caused by an acute or chronic liver disease and/or a portosystemic shunt. Its pathophysiology is still debated, although the synergic role of hyperammonemia and inflammation is now admitted for years. Several additional mechanisms have been suspected, one of them being an altered permeability of the brain blood barrier (BBB). Nevertheless, many aspects remain poorly understood.

The rise of "-omics" techniques, and especially metabolomics, allowed to identify more precisely the different metabolic pathways that are involved in the pathophysiology of HE. Using a high flow chemistry technique and multivariate data analysis, metabolomics is an accurate way to understand the pathophysiology and pathogenesis of multifactorial diseases such as HE. Several studies have been published in cirrhosis. It has been suggested that serum metabolites at admission, as well as thyroxine, can predict advanced HE in patients without brain failure. In a cohort including more than 600 patients, a higher microbially-derived metabolites, together with a lower thyroxine level, were associated with further development of brain failure. In another study from the same team, serum and urinary metabolites were significantly different in hospitalised patients who had developed poor outcome or not. Another study conducted in the CANONIC cohort as also found changes in metabolites of patients with cirrhosis and acute-on-chronic liver failure (ACLF), revealing mitochondrial dysfunction in peripheral organs that may contribute to organ failures. Last, our team previously analysed plasma and cerebrospinal fluid (CSF) samples of patients with cirrhosis and HE hospitalised in intensive care unit (ICU), showing alteration in ammonia and amino-acids metabolism, and also in energy metabolism. However, in the latest study, ALCF grading was not available. As many of these patients were in a severe condition, one could hypothesize that the metabolomic changes observed in these patients may have been confounded by an ACLF profile. Therefore, the objective of this study is to characterize the metabolomic fingerprints of HE in patients with cirrhosis, using 4 different groups of patients: patients with or without HE, with or without ALCF.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient with cirrhosis of any etiology
* Informed patient who does not object to participating in the study
* Patient affiliated to a social security scheme or entitled beneficiary

Exclusion Criteria:

* Pregnant or breast-feeding women
* Protected populations: under guardianship or trusteeship
* Previous liver transplant
* Patient on AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with cirrhosis according to the presence of ACLF or hepatic encephalopathy or not.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Metabolomic analysis by mass spectrometry from a 6mL blood sample of cirrhotic patients. | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Marika Rudler, MD, PhD, Study Chair — Sorbonne University, Pitié salpêtrière hospital
Locations (2):
- France (2):
  - Service d'hépato-gastroentérologie Hôpital Pitié Salpêtrière, Paris
  - Sorbonne University, Pitié salpêtrière hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.